CLINICAL TRIAL: NCT01081782
Title: A Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of ONO-4641 in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study of the Safety and Efficacy of ONO-4641 in Patients With Relapsing-Remitting Multiple Sclerosis
Acronym: DreaMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4641POU006
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; ONO-4641
MeSH Terms: conditions — Multiple Sclerosis | interventions — ceralifimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- E1 (Experimental)
  Interventions: Drug: ONO-4641
- E2 (Experimental)
  Interventions: Drug: ONO-4641
- E3 (Experimental)
  Interventions: Drug: ONO-4641
- P (Placebo Comparator)
  Interventions: Drug: ONO-4641 placebo

INTERVENTIONS:
Drug: ONO-4641 — 0.15 mg once per day for 26 weeks
  Arms: E1
Drug: ONO-4641 — 0.1 mg once per day for 26 weeks
  Arms: E2
Drug: ONO-4641 — 0.05 mg once per day for 26 weeks
  Arms: E3
Drug: ONO-4641 placebo — Placebo once per day for 26 weeks
  Arms: P

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ONO-4641 in patients with relapsing-remitting multiple sclerosis over a 26-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged 18-55 years inclusive at screening
* Patients who have a definite diagnosis of relapsing-remitting Multiple Sclerosis

Exclusion Criteria:

* Multiple Sclerosis course other than relapsing-remitting multiple sclerosis
* History of malignancy
* History of clinically significant chronic disease of the immune system (other than Multiple Sclerosis)
* Inability to undergo Gd-enhanced MRI scans
* Diagnosis of diabetes mellitus (type I or type II)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 407 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Total number of T-1-weighted Gd-enhanced lesions obtained with MRI at 4-week intervals for 26 weeks. | 26 weeks

SECONDARY OUTCOMES:
Total volume of Gd-enhanced lesions | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (86):
- United States (23):
  - Tucson Clinical Site 133, Tucson, Arizona
  - Aurora Clinical Site 132, Aurora, Colorado
  - Fort Collins Clinical Site 123, Fort Collins, Colorado
  - Fairfield Clinical Site 110, Fairfield, Connecticut
  - Ormond Beach Clinical Site 129, Ormond Beach, Florida
  - Sarasota Clinical Site 116, Sarasota, Florida
  - Sarasota Clinical Site 117, Sarasota, Florida
  - Northbrook Clinical Site 135, Northbrook, Illinois
  - Fort Wayne Clinical Site 111, Fort Wayne, Indiana
  - Indianapolis Clinical Site 121, Indianapolis, Indiana
  - Detroit Clinical Site 104, Detroit, Michigan
  - Farmington Hills Clinical Site 126, Farmington Hills, Michigan
  - Lebanon Clinical Site 115, Lebanon, New Hampshire
  - Albuquerque Clinical Site 106, Albuquerque, New Mexico
  - Rochester Clinical Site 108, Rochester, New York
  - Charlotte Clinical Site 125, Charlotte, North Carolina
  - HighPoint Clinical Site 128, HighPoint, North Carolina
  - Raleigh Clinical Site 103, Raleigh, North Carolina
  - Akron Clinical Site 112, Akron, Ohio
  - Philadelphia Clinical Site 120, Philadelphia, Pennsylvania
  - Knoxville Clinical Site 134, Knoxville, Tennessee
  - Round Rock Clinical Site 107, Round Rock, Texas
  - Seattle Clinical Site 118, Seattle, Washington
- Belgium (3):
  - Brugge Clinical Site 203, Bruges
  - La Louviere Clinical Site 201, La Louvière
  - Sijsele Clinical Site 202, Sijsele
- Canada (5):
  - Gatineau Clinical Site 114, Gatineau, Quebec
  - Greenfield Park Clinical Site 109, Greenfield Park, Quebec
  - Vancouver Clinical Site 131, British Columbia
  - Montreal Clinical Site 113, Québec
  - Montreal Clinical Site 102, Québec
- Czechia (4):
  - Olomouc Clinical Site 212, Olomouc
  - Ostrava Clinical Site 214, Ostrava
  - Pardubice Clinical Site 211, Pardubice
  - Praha 5 Clinical Site 213, Prague
- Germany (9):
  - Berlin Clinical Site 223, Berlin
  - Essen Clinical Site 222, Essen
  - Giessen Clinical Site 221, Giessen
  - Leipzig Clinical Site 229, Leipzig
  - Mainz Clinical Site 231, Mainz
  - Marburg Clinical Site 228, Marburg
  - Munster Clinical Site 225, Münster
  - Tubingen Clinical Site 226, Tübingen
  - Ulm Clinical Site 230, Ulm
- Greece (2):
  - Athens Clinical Site 243, Athens
  - Thessaloniki Clinical Site 245, Thessaloniki
- Japan (9):
  - Kanto Region Clinical Site 404, Kanto
  - Kanto Region Clinical Site 405, Kanto
  - Kanto Region Clinical Site 406, Kanto
  - Kanto Region Clinical Site 409, Kanto
  - Kinki Region Clinical Site 401, Kinki
  - Kinki Region Clinical Site 407, Kinki
  - Kinki Region Clinical Site 408, Kinki
  - Tohoku Region Clinical Site 403, Tōhoku
  - Tohoku Region Clinical Site 410, Tōhoku
- Poland (8):
  - Bialystok Clinical Site 305, Bialystok
  - Czeladz Clinical Site 303, Czeladź
  - Gdansk Clinical Site 302, Gdansk
  - Katowice Clinical Site 309, Katowice
  - Krakow Clinical Site 307, Krakow
  - Lodz Clinical Site 306, Lodz
  - Plewiska Clinical Site 304, Plewiska
  - Warszawa Clinical Site 308, Warsaw
- Russia (11):
  - Chelyabinsk Clinical Site 322, Chelyabinsk
  - Kaluga Clinical Site 328, Kaluga
  - Kazan Clinical Site 333, Kazan'
  - Moscow Clinical Site 332, Moscow
  - Nizhniy Novgorod Clinical Site 321, Nizhny Novgorod
  - Novosibirsk Clinical Site 324, Novosibirsk
  - St. Petersburg Clinical Site 325, Saint Petersburg
  - St. Petersburg Clinical Site 327, Saint Petersburg
  - Samara Clinical Site 328, Samara
  - Ufa Clinical Site 326, Ufa
  - Yaroslavl Clinical Site 331, Yaroslavl
- Spain (6):
  - Barcelona Clinical Site 252, Barcelona
  - Barcelona Clinical Site 253, Barcelona
  - Bilbao Clinical Site 255, Bilbao
  - Girona Clinical Site 254, Girona
  - Hospitalet de Llobregat Clinical Site 251, L'Hospitalet de Llobregat
  - Sevilla Clinical Site 256, Seville
- Ukraine (6):
  - Dnipropetrovsk Clinical Site 341, Dnipropetrovsk
  - Donetsk Clinical Site 345, Donetsk
  - Kharkiv Clinical Site 346, Kharkiv
  - Kyiv Clinical Site 344, Kyiv
  - Lviv Clinical Site 343, Lviv
  - Vinnytsya Clinical Site 342, Vinnytsia